CLINICAL TRIAL: NCT00927407
Title: A Randomized, Single-Dose, Parallel Group, Comparative Pharmacokinetic (PK) Study to Evaluate Malathion Gel 0.5% Versus Ovide (Malathion) Lotion 0.5% in Patients With Pediculosis Capitis
Brief Title: Pharmacokinetics of Malathion Gel 0.5% and Malathion 0.5% Lotion (Ovide) in Patients With Head Lice
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MALG-0603
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Pediculosis
Keywords: Head Lice
MeSH Terms: conditions — Lice Infestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Malathion gel 0.05% (Experimental): Malathion gel 0.5% topical treatment for head lice
  Interventions: Drug: Malathion gel 0.5%
- Malathion lotion 0.5% (Active Comparator): Malathion lotion 0.5% treatment for head lice
  Interventions: Drug: Malathion lotion 0.5%

INTERVENTIONS:
Drug: Malathion gel 0.5% — Malathion gel 0.5% applied to the scalp for 30 minutes
  Other Names: MALG
  Arms: Malathion gel 0.05%
Drug: Malathion lotion 0.5% — Malathion lotion 0.5% applied to scalp for 12 hours
  Other Names: OVIDE lotion
  Arms: Malathion lotion 0.5%

SUMMARY:
In this study, 24 adult patients with head lice will be treated with a topical malathion head lice treatment; 12 patients will be treated with a novel product, Malathion Gel, 0.5%, and other 12 patients will be treated with Ovide Lotion 0.5% marketed by Taro Pharmaceuticals USA, Inc. The primary objective of this study is to compare the blood level exposure of Malathion 0.5% Gel to that of the OVIDE Lotion 0.5%.

DETAILED DESCRIPTION:
A randomized, single-dose, parallel group, comparative PK study. Patients will be randomly assigned in 1:1 ratio to the study products. Twenty four (24) consenting patients, age 18 years and older, who meet Inclusion/Exclusion criteria will be enrolled in this study. 12 Patients will be treated with Malathion Gel, 0.5% and other 12 Patients will be treated with Ovide Lotion 0.5%. The study will be single centre and conducted only in India. The primary objective of this study is to compare the systemic exposure of Malathion 0.5% Gel manufactured by Taro Pharmaceuticals USA, Inc. to that of the OVIDE Lotion 0.5%, currently marketed by Taro Pharmaceutical USA, Inc., in adult Patients with head lice. The secondary objective is to determine the link between the exposure and cholinesterase activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female
* Patients 18 years of age or older and healthy presenting with Pediculosis capitis
* The Patient must be willing to consent to the Patient's treatment with Malathion Gel 0.5% or Ovide Lotion 0.5% and for blood drawings before and after medication administration.

Exclusion Criteria:

* Individuals with history of irritation or sensitivity to pediculicides or hair care products
* Individuals with any visible skin/scalp condition at the treatment site which, in the opinion of the investigative personnel, or Sponsor, will interfere with the evaluation.
* Individuals previously treated with a pediculicide within 4 weeks of the study.
* Individuals who exhibit potential signs and symptoms of cholinesterase inhibition.
* Patients currently receiving sulfonamide antibiotics or ivermectin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Measurement of blood and urinary levels of malathion and metabolites | 48 hours

SECONDARY OUTCOMES:
Measure cholinesterase levels and compare to malathion metabolite levels | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator Site, Rabale, Navi Mumbai, India

REFERENCES:
- [Background] Meinking TL, Vicaria M, Eyerdam DH, Villar ME, Reyna S, Suarez G. A randomized, investigator-blinded, time-ranging study of the comparative efficacy of 0.5% malathion gel versus Ovide Lotion (0.5% malathion) or Nix Creme Rinse (1% permethrin) used as labeled, for the treatment of head lice. Pediatr Dermatol. 2007 Jul-Aug;24(4):405-11. doi: 10.1111/j.1525-1470.2007.00460.x. PMID 17845167